CLINICAL TRIAL: NCT00549601
Title: A Multi-center, Randomised, Open-label Study to Evaluate Convenience and Safety of Change in the Mode of Administration of Rivastigmine (From Capsules to a Transdermal Patch) in Patients With Alzheimer's Disease
Brief Title: Convenience, Tolerability, and Safety of Change in the Administration of Rivastigmine From Capsules to a Transdermal Patch in Patients With Mild to Moderate Alzheimer's Disease
Acronym: KAPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CENA713DES07
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's; rivastigmine; transdermal; safety; randomized; switch; patch
MeSH Terms: conditions — Alzheimer Disease | interventions — Rivastigmine

ARMS (3):
- Rivastigmine patch (4.6 mg/day switch to 9.5 mg/day) (Experimental)
  Interventions: Drug: Rivastigmine patch (4.6 mg/day switch to 9.5 mg/day)
- Rivastigmine patch (9.5 mg/day) (Experimental)
  Interventions: Drug: Rivastigmine patch (9.5 mg/day)
- Rivastigmine capsules (6 mg to 12 mg/day) (Active Comparator)
  Interventions: Drug: Rivastigmine capsules (6 mg to 12 mg/day)

INTERVENTIONS:
Drug: Rivastigmine patch (4.6 mg/day switch to 9.5 mg/day) — Rivastigmine administered transdermally via patches at increasing doses (1 patch/day of 4.6 mg for the first month, changing to 1 patch/day of 9.5 mg for the remaining two months).
  Arms: Rivastigmine patch (4.6 mg/day switch to 9.5 mg/day)
Drug: Rivastigmine patch (9.5 mg/day) — Rivastigmine administered transdermally via patches at a constant dose (9.5 mg/day for the 3 months of treatment).
  Arms: Rivastigmine patch (9.5 mg/day)
Drug: Rivastigmine capsules (6 mg to 12 mg/day) — Rivastigmine administered orally, following the same regime as prior to randomization (doses between 6 mg and 12 mg/day), which remained unchanged throughout the 3 months of treatment.
  Arms: Rivastigmine capsules (6 mg to 12 mg/day)

SUMMARY:
This study used two doses of rivastigmine transdermal patch (5 cm^2, 10 cm^2) to establish the feasibility of 2 switch schedules (with transdermal patch one-step dose titration or without dose titration) from rivastigmine capsules (3 mg bid (bis in die, twice a day), 4,5 mg bid, 6 mg bid) to rivastigmine transdermal patch and to assess safety, tolerability, convenience, and caregivers preferences of rivastigmine transdermal patch versus capsules.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV (Diagnostic & Statistical Manual of Mental Disorders, Version IV) criteria for dementia of Alzheimer type and NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association) criteria for probable Alzheimer's disease (AD), have a MMSE (Mini Mental State Examination) score > 10 and < 26
* Have received continuous treatment with rivastigmine capsules at least with 3 mg bid (6 mg of total daily dose) for at least 3 months before entering in the study
* Cooperative, willing to complete all aspects of the study, and capable of doing so, either alone or with the aid of a responsible caregiver
* Have a primary caregiver willing to accept responsibility for supervising the treatment, (eg, application and removal of the patch daily at approximately the same time of day) and assessing the condition of the patient throughout the study.

Exclusion Criteria:

* A medical or neurological condition other that AD that could explain the patients dementia (eg, Huntington's disease, Parkinson's Disease, abnormal thyroid function test, B12 or folate deficiency, post-traumatic conditions, syphilis)
* Current diagnosis of an active skin lesion/disorder that would prevent accurate assessment of the adhesion and potential skin irritation of the patch (e.g., atopic dermatitis, wounded or scratched skin in the area of the patch application)
* History of allergy to topical products containing vitamin E
* Taken any of the following substances prior to randomization:

  * succinylcholine-type muscle relaxants during the previous 2 weeks
  * an investigational drug during the previous 4 weeks

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, MD, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Period: Randomized
Arm/Group | Rivastigmine Patch (4.6 mg/Day Switch to 9.5 mg/Day) | Rivastigmine Patch (9.5 mg/Day) | Rivastigmine Capsules (6 mg to 12 mg/Day)
Started | 43 | 48 | 51
Completed | 43 | 47 | 49
Not Completed | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Period: Received Study Drug
Arm/Group | Rivastigmine Patch (4.6 mg/Day Switch to 9.5 mg/Day) | Rivastigmine Patch (9.5 mg/Day) | Rivastigmine Capsules (6 mg to 12 mg/Day)
Started | 43 (Subjects who started this period (safety population) received at least 1 dose of study drug.) | 47 (Subjects who started this period (safety population) received at least 1 dose of study drug.) | 49 (Subjects who started this period (safety population) received at least 1 dose of study drug.)
Completed | 36 | 36 | 45
Not Completed | 7 | 11 | 4
Not completed — Adverse Event | 2 | 5 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Protocol Violation | 3 | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivastigmine Patch (4.6 mg/Day Switch to 9.5 mg/Day) | Rivastigmine Patch (9.5 mg/Day) | Rivastigmine Capsules (6 mg to 12 mg/Day) | Total
Number analyzed (Participants) | 43 | 47 | 49 | 139
Age Continuous [Mean (Standard Deviation); unit: years] | 77.05 (4.82) | 75.34 (7.25) | 77.35 (6.62) | 76.58 (6.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 25 | 84
  Male | 13 | 18 | 24 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Had a Gastrointestinal Adverse Event (AE) at Any Time During the Study
Description: Gastrointestinal adverse events (including nausea, vomiting, and diarrhea) were coded using the medical dictionary MedDRA v11.0 and the number of patients who suffered an AE were described by system organ class (SOC) and preferred term (PT).
Time Frame: Baseline to end of study (Month 3)
Population: The Safety population included all randomized patients who received at least one dose of the study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivastigmine Patch (4.6 mg/Day Switch to 9.5 mg/Day) | Rivastigmine Patch (9.5 mg/Day) | Rivastigmine Capsules (6 mg to 12 mg/Day)
Number analyzed (Participants) | 43 | 47 | 49
Percentage of participants | 4.65 (4.65) | 4.26 (4.26) | 6.12 (6.12)

2. Secondary Outcome: Percentage of Patients With an AE Involving the Skin (Local Tolerance) Recorded Over the Course of the Study Period (Patch Groups Only)
Description: Adverse events involving the skin included urticaria, pruritus, erythema, and pigmentation disorder. Only the groups administered rivastigmine transdermally via patch were analyzed. The adverse events were coded using the medical dictionary MedDRA v11.0 and the number of patients who suffered an AE were described by system organ class (SOC) and preferred term (PT).
Time Frame: Baseline to end of study (Month 3)
Population: The Safety population included all randomized patients who received at least one dose of the study medication.
Measure: Number; unit: Percentage of participants
Groups:
- Rivastigmine 4.6 mg/9.5 mg Patch: Rivastigmine transdermal patches at increasing doses: Application of one 4.6 mg patch every day for the first month of treatment and thereafter daily application of one 9.5 mg patch for the next two months.
- Rivastigmine 9.5 mg Patch: Rivastigmine transdermal patches at a constant dose: Application of one 9.5 mg patch every day for the whole treatment period.
Arm/Group | Rivastigmine 4.6 mg/9.5 mg Patch | Rivastigmine 9.5 mg Patch
Number analyzed (Participants) | 43 | 47
Percentage of participants | 11.63 (11.63) | 17.02 (17.02)

3. Secondary Outcome: Percentage of Patients With at Least 1 AE of Any Kind Recorded During the Period of the Study.
Description: Adverse events were coded using the medical dictionary MedDRA v11.0 and the number of patients who suffered an AE were described by system organ class (SOC) and preferred term (PT). They were also tabulated by severity, relationship with study treatment, and action taken.
Time Frame: Baseline to end of study (Month 3)
Population: The Safety population included all randomized patients who received at least one dose of the study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivastigmine Patch (4.6 mg/Day Switch to 9.5 mg/Day) | Rivastigmine Patch (9.5 mg/Day) | Rivastigmine Capsules (6 mg to 12 mg/Day)
Number analyzed (Participants) | 43 | 47 | 49
Percentage of participants | 48.84 (48.84) | 55.32 (55.32) | 53.06 (53.06)

4. Secondary Outcome: Overall Caregiver Satisfaction With Treatment
Description: Caregivers were asked to rate their overall degree of satisfaction with the Alzheimer's disease treatment on a scale of 1 to 5 (1 "Very good" - 5 "Very poor") at the end of the study (Month 3). A higher score indicates less satisfaction.
Time Frame: At end of study (Month 3)
Population: The Safety population included all randomized patients who received at least one dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Rivastigmine Patch (4.6 mg/Day Switch to 9.5 mg/Day) | Rivastigmine Patch (9.5 mg/Day) | Rivastigmine Capsules (6 mg to 12 mg/Day)
Number analyzed (Participants) | 43 | 47 | 49
Participants
  Not Decided (ND) | 1 | 3 | 1
  Very good | 18 | 20 | 10
  Good | 18 | 14 | 33
  Average | 3 | 5 | 2
  Poor | 3 | 2 | 3
  Very Poor | 0 | 3 | 0

5. Secondary Outcome: Overall Patient Satisfaction With Treatment
Description: Patients were asked to rate their overall degree of satisfaction with the Alzheimer's disease treatment on a scale of 1 to 5 (1 "Very good" - 5 "Very poor") at the end of the study (Month 3). A higher score indicates less satisfaction.
Time Frame: At end of study (Month 3)
Population: The Safety population included all randomized patients who received at least one dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Rivastigmine Patch (4.6 mg/Day Switch to 9.5 mg/Day) | Rivastigmine Patch (9.5 mg/Day) | Rivastigmine Capsules (6 mg to 12 mg/Day)
Number analyzed (Participants) | 43 | 47 | 49
Participants
  Not Decided (ND) | 0 | 3 | 1
  Very good | 18 | 14 | 12
  Good | 20 | 21 | 29
  Average | 3 | 6 | 5
  Poor | 2 | 2 | 2
  Very Poor | 0 | 1 | 0

6. Secondary Outcome: Change in the Total Mini-Mental State Examination (MMSE) Score From Baseline to Month 1 and Month 3
Description: The Mini Mental State Examination (MMSE) was used to evaluate the patient's cognitive status and how it progressed over time. The 35-point version used in this study was made up of five sections: orientation, fixation, attention and calculation, memory and language, and constructional praxis. The total score for each patient was obtained by adding the score from each of the above sections. The individual receives 1 point for each correct answer. The total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement.
Time Frame: Baseline to Month 1 and Month 3
Population: The Safety population was made up of all the randomized patients who had taken at least one dose of the study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rivastigmine Patch (4.6 mg/Day Switch to 9.5 mg/Day) | Rivastigmine Patch (9.5 mg/Day) | Rivastigmine Capsules (6 mg to 12 mg/Day)
Number analyzed (Participants) | 43 | 47 | 49
Units on a scale
  Month 1 | 0.12 (2.60) | 0.59 (2.58) | 1.00 (2.63)
  Month 3 | -0.59 (2.85) | 0.12 (2.85) | -0.40 (2.42)

ADVERSE EVENTS:
Arm/Group | Rivastigmine Patch (4.6 mg/Day Switch to 9.5 mg/Day) | Rivastigmine Patch (9.5 mg/Day) | Rivastigmine Capsules (6 mg to 12 mg/Day)
Serious Adverse Events (participants affected / at risk) | 2/43 | 3/47 | 1/49
Other Adverse Events (participants affected / at risk) | 8/43 | 7/47 | 8/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine Patch (4.6 mg/Day Switch to 9.5 mg/Day) (N=43) | Rivastigmine Patch (9.5 mg/Day) (N=47) | Rivastigmine Capsules (6 mg to 12 mg/Day) (N=49)
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cerebellar haematoma (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine Patch (4.6 mg/Day Switch to 9.5 mg/Day) (N=43) | Rivastigmine Patch (9.5 mg/Day) (N=47) | Rivastigmine Capsules (6 mg to 12 mg/Day) (N=49)
Application site erythema (General disorders) | 3 | 5 | 0
Application site pruritus (General disorders) | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 6
Agitation (Psychiatric disorders) | 3 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.